DMID 16-0095 Protocol Version Date: 3/22/2019

# **CONSENT FORM**

UAB IRB Approved 22-May-2019 until 21-May-2020

TITLE OF RESEARCH: A Phase II, Single-Stage, Single-Arm Investigation of Oral Valganciclovir

Therapy in Infants with Asymptomatic Congenital Cytomegalovirus

Infection

**SCREENING CONSENT** 

IRB PROTOCOL NO.: IRB-300001001

INVESTIGATOR: David Kimberlin, MD

**SPONSOR:** National Institutes of Allergy and Infectious Disease and Genetech, Inc.

SPONSOR PROTOCOL NO.: DMID 16-0095

# **Purpose of the Research**

| General Information | You are being asked to take part in a research study. This research study is |
|---|---|
| | voluntary, meaning you do not have to take part in it. The procedures, risks, and |
| | benefits are fully described further in the consent form. |
| Purpose | The purpose of the study is to evaluate if treatment with an approved drug |
| | called Valganciclovir, will reduce the risk of hearing loss developing in babies |
| | with Congenital CMV, but have no symptoms at birth. |
| Duration & Visits | You will be in this portion of the study for less than 30 days. We will swab your |
| | baby's mouth and if the results are positive, we will schedule your baby to have |
| | a second swab, a urine specimen collection and a hearing test done. |
| Overview of Procedures | If your baby's first swab of their mouth is positive a second mouth swab and a |
| | urine specimen will be collected will be done to confirm the test results. Both |
| | CMV tests are done by a simple cheek swab. The urine specimen will be |
| | collected by way of cotton balls in diaper or from a urine collection bag. |
| | This phase of the study will include 2 mouth swabs and a urine collection. |
| | hearing evaluation. |
| Risks | The mouth swab and the urine collection should not cause discomfort to |
| | your baby. There are no risks associated with these procedures. |
| Benefits | The benefit to you for participation in this study is that you will find out if your |
| | baby does or does not have a congenital CMV infection. If your baby is positive |
| | for congenital CMV infection you will be given the opportunity to participate in |
| | our treatment study. |
| Alternatives | The alternative is to not participate in this screening for CMV. The study doctor |
| | will be available to discuss with you the alternatives to your baby's participation and their risks and benefits. |

Protocol Version Date: 3/22/19

You are being asked to allow your baby to participate in a research study of cytomegalovirus infection. Cytomegalovirus (CMV) is the leading cause of congenital infection - infection of the baby while it is still in the mother's womb. It is estimated that 5 to 10 out of every 1000 babies born will have a congenital CMV infection. Although most babies with congenital CMV infection do not have any problems due to the virus, around 15% will have hearing loss, visual problems, physical or developmental disabilities. The hearing loss due to congenital CMV infection can be present at birth or can develop later during childhood. Overall Congenital CMV is a rare infection at birth, but it accounts for 21% of hearing loss at birth and 24% of hearing loss by age 4.

This study is being done to evaluate if treatment with an approved drug called Valganciclovir, will reduce the risk of hearing loss developing in babies with Congenital CMV, but have no symptoms at birth.

We are screening newborns at UAB for CMV, to identify those who are born with CMV infection, but show no outward symptoms.

## **Study Participation and Procedures**

In this study, we plan to screen approximately 48,250 newborns at all study sites across the USA We plan to screen approximately 5361 newborns at this site to identify eligible subjects (those with a positive CMV screening test). If your baby's screening test is positive a second test will be done to confirm the test results. Both CMV tests are done by a simple cheek swab at no cost to you, but with your consent. The study doctor will discuss with you your responsibilities as a participant.

If you allow your baby to participate in this study, we will start by obtaining consent to participate. We will then test to see if your baby has CMV. Your participation will include filling out the contact form with your name, address, phone number and demographics such as date of birth and race. We will ask you to sign a form allowing us to access your UAB medical records to gather information for the study such as the hearing assessment or other interventions for the baby or for you.

- If your baby's CMV test is **negative** in the screening phase of the study, your participation is complete. There is no further study related activity or involvement.
- If your baby's initial screening CMV test is **positive**:
  - 1. We will schedule a second CMV test and urine collection to confirm the results.
  - 2. We will give you a urine collection kit containing cotton balls and instructions which you can use prior to returning to us for the second confirmatory test.
  - 3. We will schedule your baby for a complete hearing exam.
  - 4. We will also obtain the results of your baby's newborn hearing test done at UAB.

If your baby is positive for a congenital CMV infection, you will be contacted regarding recommendation for follow up for CMV. We will also discuss your options to allow your baby to participate in the treatment study with Valganciclovir. If you decide to allow your baby to participate in the treatment portion of this study, another informed consent will be presented


Protocol Version Date: 3/22/19

and discussed in detail. We plan to give you the information and will send a letter informing your pediatrician of the diagnosis at your request.

### **Risks and Discomforts**

### Saliva Collection:

Your baby will have the inside of his/her cheek swabbed to collect a saliva sample. This should not be uncomfortable for your baby. And there are no associated risks with this procedure.

## **Urine Collection:**

Your baby will have cotton balls placed in his/her diaper and we will obtain the urine from those cotton balls or a urine bag placed over his/her genitals once you return to the CHRU for the second confirmatory oral swab. There are no associated risks with this procedure other than slight redness where the urine bag is attached to the skin. We will give you a kit containing cotton balls and instructions to use in case of a positive CMV oral swab.

### **Benefits**

The benefit to you for participation in this study is that you will find out if your baby does or does not have a congenital CMV infection. If your baby is positive for congenital CMV infection you will be given the opportunity to participate in our treatment study.

### **Alternatives**

The alternative is to not participate in this screening for CMV. The study doctor can be available to discuss with you the alternatives to your baby's participation and their risks and benefits.

### Confidentiality

Federal regulations give you certain rights related to your baby's health information. These include the right to know who will be able to get the information and why they may be able to get it. The study doctor must get your authorization (permission) to use or give out any health information that might identify your baby. The information obtained about your baby for this study will be kept confidential to the extent allowed by law. Your baby's personal information will be kept secure in a locked file and all other data will be secure on a database as well as coded by a number and not your baby's name or personal information. Some of your baby's information may be transmitted electronically (by email or by fax) but it will be coded to assure confidentiality. A copy of your baby's consent form will be placed in your baby's medical record at Children's Hospital

Therefore, research information that identifies your baby may be shared with the UAB Institutional Review Board (IRB) and others who are responsible for ensuring compliance with laws and regulations related to research, including people on behalf of your baby's doctor and the research study team, and the FDA according to regulation 21 CFR 50.25(a(5).

Monitors, auditors, the Institutional Review Board for Human Use, and regulatory authorities will be


Protocol Version Date: 3/22/19

granted direct access to your original medical records for verification of trial procedures and/or data without violating confidentiality.

Data and samples collected for this study will use a study ID # as a unique identifier. There is a minimal risk of a break in confidentiality.

# What protected health information may be used and/or given to others?

All medical information, including but not limited to information and/or records of any diagnosis or treatment of disease or condition, which may include sexually transmitted diseases (e.g., HIV, etc.) or communicable diseases, drug/alcohol dependency, etc.; all personal identifiers, including but not limited to your name, social security number, medical record number, date of birth, dates of service, etc.; any past, present, and future history, examinations, laboratory results, imaging studies and reports and treatments of any kind, including but not limited to drug/alcohol treatment, psychiatric/psychological treatment; financial/billing information, including but not limited to copies of your medical bills; any other information related to or collected for use in the research study, regardless of whether the information was collected for research or non-research (e.g., treatment) purposes; records about any study drug you received or about study devices used; and consent forms from past studies that might be in your baby's medical record.

Your baby's consent form will be placed in your baby's medical record at UAB Health System or Children's of Alabama. This may include either a paper medical record or electronic medical record (EMR). An EMR is an electronic version of a paper medical record of your baby's care within this health system. Your baby's EMR may indicate that your baby is on a clinical trial and provide the name and contact information for the principal investigator.

If your baby is receiving care or has received care within this health system (outpatient or inpatient) and is participating in a research study, results of research tests or procedures (i.e. laboratory tests, imaging studies and clinical procedures) may be placed in your baby's existing medical record.

If your baby has never received care within this health system (outpatient or inpatient) and is participating in a research study, a medical record will be created for your baby to maintain results of research tests or procedures.

Results of research tests or procedures may be placed in your baby's medical record. All information within your baby's medical record can be viewed by individuals authorized to access the record.

Information relating to this study, including your baby's name, medical record number, date of birth and social security number, may be shared with the billing offices of UAB and UAB Health System affiliated entities, along with Children's of Alabama and its billing agents so costs for clinical services can be appropriately paid for by either the study account or by your insurance.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify your baby. At most, the Web site will include a summary of the results. You can search this Web site at any time.


Protocol Version Date: 3/22/19

# Who may use and give out information about you?

Information about your health may be used and given to others by the study doctor and staff. They might see the research information during and after the study.

# Who might get this information?

All Individuals/entities listed in the informed consent document(s), including but not limited to, the physicians, nurses and staff and others performing services related to the research (whether at UAB or elsewhere). Your information may also be given to the sponsor of this research. "Sponsor" includes any persons or companies that are working for or with the sponsor, or are owned by the sponsor, or are providing support to the sponsor (e.g., contract research organization).

Information about you and your health which might identify you may be given to:

- the Office for Human Research Protections (OHRP)
- the U.S. Food and Drug Administration (FDA)
- Department of Health and Human Services (DHHS) agencies
- Governmental agencies in other countries
- Governmental agencies to whom certain diseases (reportable diseases) must be reported
- the University of Alabama at Birmingham the physicians, nurses and staff working on the research study (whether at UAB or elsewhere); other operating units of UAB, UAB Hospital, UAB Highlands Hospital, University of Alabama Health Services Foundation, Children's of Alabama, Eye Foundation Hospital, and the Jefferson County Department of Health, as necessary for their operations; the UAB IRB and its staff
- the billing offices of UAB and UAB Health Systems affiliates and/or Children's of Alabama and its billing agents

## Why will this information be used and/or given to others?

Information about you and your health that might identify you may be given to others to carry out the research study. The sponsor will analyze and evaluate the results of the study. In addition, people from the sponsor and its consultants will be visiting the research site. They will follow how the study is done, and they will be reviewing your information for this purpose.

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. The researchers may not disclose or use your baby's information, documents, or specimens that may identify your baby in any federal, state, or local civil, criminal, administrative, legislative, or other action such as a suit or other proceeding without your consent. If there is a court subpoena, information, documents or specimens collected about your baby as part of this study cannot be disclosed to anyone else who is not connected with the research, except if there is a law that requires disclosure (such as to report child abuse or a communicable disease). This certificate does not prohibit requests for information from the groups listed above, who are responsible for overseeing the study.

The Certificate cannot be used to refuse a request for information from personnel of the United States federal or state government agency sponsoring the project that is needed for auditing or program evaluation by the *National Institutes of Health* which is funding this project or for information that must be disclosed in order to meet the requirements of the federal Food and Drug Administration (FDA). You should understand that a Certificate of Confidentiality does not prevent

IC Version Date: 05/15/19


#### Protocol Version Date: 3/22/19

you from voluntarily releasing information about yourself or your involvement in this research. If you want your research information released to an insurer, medical care provider, or any other person not connected with the research, you must provide consent to allow the researchers to release it.

The Certificate of Confidentiality will not be used to prevent disclosure for any purpose you have consented to in this informed consent document.

### What if I decide not to give permission to use and give out my health information?

By signing this consent form, you are giving permission to use and give out the health information listed above for the purposes described above. If you refuse to give permission, you will not be able to be in this research.

# May I review or copy the information obtained from me or created about me?

You have the right to review and copy your health information. However, if you decide to be in this study and sign this permission form, you will not be allowed to look at or copy your information until after the research is completed.

# May I withdraw or revoke (cancel) my permission?

Yes, but this permission will not stop automatically. The use of your personal health information will continue until you cancel your permission.

You may withdraw or take away your permission to use and disclose your health information at any time. You do this by sending written notice to the study doctor. If you withdraw your permission, you will not be able to continue being in this study.

When you withdraw your permission, no new health information which might identify you will be gathered after that date. Information that has already been gathered may still be used and given to others. This would be done if it were necessary for the research to be reliable.

## Is my health information protected after it has been given to others?

If you give permission to give your identifiable health information to a person or business, the information may no longer be protected. There is a risk that your information will be released to others. Including others outside of UAB, without your permission.

## **Voluntary Participation and Withdrawal**

Whether or not you allow your baby to take part in this study is your choice. There will be no penalty if you decide to withdraw your baby from the study. If you decide not to allow your baby to be in the study, you will not lose any benefits otherwise owed. You are free to withdraw your baby from this research study at any time. Your choice to withdraw your baby from the study will not affect your baby's relationship with this institution.


Protocol Version Date: 3/22/19

Your baby may be removed from the study without your consent if the sponsor ends the study, or if for any other reasons in the opinions of both the site investigator as well as the study chairperson, that ending study participation is the best course of action for your baby.

# **Cost of Participation**

There will be no cost to your baby for taking part in this study.

The costs of your baby's standard medical care will be billed to you and/or your insurance company in the usual manner.

# **Payment for Participation in Research**

The study will provide a small gift as a token of appreciation (valued approximately \$10) at the time of the initial screening. If your baby's initial test is positive for Congenital CMV, you will be asked to return for a second screening. After you complete the second screening and hearing test, you will be paid \$25. Ask the study staff about the method of payment that will be used for this study (e.g., check, cash, gift card, direct deposit).

## **Payment for Research-Related Injuries**

UAB, Genentech and the sponsor (National Institutes of Health), have not provided for any payment if your baby is harmed as a result of taking part in this study. If such harm occurs, treatment will be provided. However, this treatment will not be provided free of charge.

## **Significant New Findings**

You will be told by doctor or the study staff if any new information becomes available that might affect your choice to stay keep your baby in the study.

### Questions

If you have any questions, concerns, or complaints about the research or a research-related injury including available treatments, please contact the research doctor, Dr. Kimberlin will be glad to answer any of your questions. Dr. Kimberlin's number is 205-934-2424. Dr. Kimberlin may also be reached after hours by paging him at 205-934-3411.

If you have questions about your baby's rights as a research participant, or concerns or complaints about the research, you may contact the UAB Office of the IRB (OIRB) at (205) 934-3789 or toll free at 1-855-860-3789. Regular hours for the OIRB are 8:00 a.m. to 5:00 p.m. CT, Monday through Friday. You may also call this number in the event the research staff cannot be reached or you wish to talk to someone else.


You are not waiving any of your baby's legal rights by signing this informed consent document.


# **Storage of Specimens for Future Use**

Some specimens obtained from your baby during this study will be stored indefinitely in laboratories at the University of Alabama at Birmingham (UAB) and may be used in future virus research at UAB and at other laboratories. These specimens will be labeled with a code number that can be linked to your baby but will not include your baby's name. Any additional research studies beyond the current study using your baby's identifiable samples/cultures will be reviewed by the investigator's Institutional Review Board (IRB), a special committee that oversees medical research studies to protect the rights and welfare of the human subject volunteers. There will be no human genetic tests performed on your baby's samples/cultures.

All results from future studies using your baby's specimens will be included in the study records. No results from these studies will be placed in your baby's medical records.

| results from these studies will be placed in your baby's medical rec | ords. |
|---|---|
| Please indicate whether you will permit your baby's specimens to initialing one of the following statements: | pe used in future virus research by |
| I agree to allow my baby's specimens to be preserved f | or future virus research. |
| I do not agree to allow my baby's specimens to be pres | erved for future virus research. |
| If, in the future, you decide that you do not want your baby's special please notify Dr. Kimberlin or the Study RN at this number 205-934 1600 7th Avenue South, CHB 303, Birmingham, Al 35233, and your | -2424, or in writing at this address, |
| If you decide that you do not want your baby's specimens used for future virus research, your baby may still participate in the study. Your baby's specimens will be destroyed once all study tests are completed. | |
| Signatures | |
| You are making a decision whether or not to have your baby participates that you have read (or have been read) the information pallow your baby to participate. You will receive a copy of this signs | rovided above and decided to |
| , | /child/minor) was waived because |
| of age. | |
| Signature of Parent or Guardian | Date |
| Signature of Parent or Guardian | Date |


| DMID 16-0095 Protocol Version Date: 3/22/19 | |
|-----------------------------------------------------------------|----------|
| Signature of Principal Investigator or Person Obtaining Consent | <br>Date |

 IC Version Date: 05/15/19